CLINICAL TRIAL: NCT03061682
Title: Implantation of Add on Lens for Age Related Macular Degeneration Patients With Low Vision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, rita ehrlich, Principal Investigator, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0408-15RMC
Record Dates: First submitted 2016-12-01; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Inclusion Criteria

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Add on lens (Experimental)
  Interventions: Device: "Scharioth" macula lens A45sml/A45smy

INTERVENTIONS:
Device: "Scharioth" macula lens A45sml/A45smy — Implantation of an add on intraocular lens to low vision patients

SUMMARY:
Age related macular degeneration (AMD) is the leading cause of vision loss in patients older than 55 years old. AMD can present as dry AMD or wet AMD. In most cases AMD affects both eyes although in many cases it's asymmetrical as far as severity. Some patients require low vision aids to continue their daily life tasks. In the past a few attempts were made to use low vision intraocular lenses with corrective glasses without enough success. In addition telescopic and prismatic lenses were also tried. The difficulties with these lenses included low field of vision, unsatisfactory magnification, complicated surgical technique and high complication rates.

Recently an add on lens was designed for the sulcus for implantation in pseudophakic AMD patients. The add on lens doubles the magnification of the central image dependent on the reading distance and the anatomy of the eye.

The lens is acrylic hydrophobic and designed for implantation in the sulcus either in pseudophakic patients or in addition to an intraocular lens implanted during a routine cataract surgery. The lens is 13 mm wide with 4 symmetric haptics. The lens has 1.5 mm central part of 10 diopters and the rest of the lens has no optical power.

Our purpose is to study implantation of the lenses in AMD patients to improve their reading ability and to improve their daily living.

DETAILED DESCRIPTION:
Study design Prospective study on implantation of the add on lenses in AMD patients. The study was approved by Rabin medical center IRB.

Patients will be examined for best corrected visual acuity prior to the surgery at 6 meter and for reading at 40 and 15 cm. Improvement of the reading ability at 15 cm compared to 40 cm will predict the potential for vision improvement with the add on lens.

Before the surgery patients will have a full ophthalmological examination. Patients will have axial length and keratometry examination using the biometry. The lens will be implanted in surgery through a 2.2 mm clear cornea and will be injected and positioned in the sulcus.

Patients will be followed up at 1 day, 1 week, 4 weeks, 4 and 6 months following surgery. During follow up patients will undergo full ophthalmic exam and well as visual acuity both for distance and near.

ELIGIBILITY:
Inclusion Criteria:

* Pseudophakic patients with non-active AMD that complain on near distance reading with a distance visual acuity better than 6/60.

Exclusion Criteria:

* Exudative AMD with fluids, advanced glaucoma, advance visual field defects, aphakia, following complicated cataract surgery with PCIOL in the sulcus , phacodonesis, chronic uveitis, rubeosis iridis, central corneal opacity.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
near visual acuity | last study visit - 6 months post surgery